CLINICAL TRIAL: NCT02918331
Title: A Phase 1b Study of JNJ-54767414 (Daratumumab) in Combination With Lenalidomide and Dexamethasone (DRd) in Japanese Subjects With Previously Untreated Multiple Myeloma Who Are Ineligible for High-dose Therapy and Autologous Stem Cell Transplantation
Brief Title: A Study of JNJ-54767414 (Daratumumab) in Combination With Lenalidomide and Dexamethasone in Japanese Participants With Previously Untreated Multiple Myeloma Who Are Ineligible for High-dose Therapy and Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108197; 54767414MMY1006 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab with Lenalidomide and dexamethasone (Experimental): Daratumumab (16 milligram per kilogram [mg/kg]) will be administered by intravenous [IV] infusion to all participants once every week for 8 weeks; then once every other week for 16 weeks; thereafter once every 4 weeks until documented progression, unacceptable toxicity or study end.
  Participants will receive lenalidomide 25 mg orally on Days 1 through 21 of each 28 day cycle.
  Participants will receive dexamethasone 40mg weekly, at day 1, 8, 15, 22 of each cycle.
  Interventions: Drug: Daratumumab (16 mg/kg); Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab (16 mg/kg) — Daratumumab (16 mg/kg) will be administered by IV infusion to all participants once every week for 8 weeks; then once every other week for 16 weeks; thereafter once every 4 weeks until documented progression, unacceptable toxicity or study end.
Drug: Lenalidomide — Participants will receive lenalidomide 25 mg orally on Days 1 through 21 of each 28 day cycle. Participants with creatinine clearance (CrCl) between 30 and 60 milliLitre (mL)/minute (min) will receive lenalidomide 10 mg every 24 hours.
Drug: Dexamethasone — Participants will receive dexamethasone 40 mg weekly, at day 1, 8, 15, 22 of each cycle.

SUMMARY:
The purpose of this study is to evaluate the safety of daratumumab when combined with lenalidomide and dexamethasone in Japanese participants with newly diagnosed multiple myeloma who are not candidates for high-dose chemotherapy and autologous stem cell transplantation (ASCT).

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented multiple myeloma (MM) satisfying the CRAB (calcium elevation, renal insufficiency, anemia, and bone abnormalities) criteria , monoclonal plasma cells in the bone marrow more than equal to (>=) 10 percent (%) or presence of a biopsy proven plasmacytoma, and measurable disease Measurable disease as defined by any of the following: (a) immunoglobulin (Ig) G MM: serum monoclonal paraprotein (M protein) level >=1.0 gram/deciliter (dL) or urine M protein level >= 200 milligram(mg)/24 hours; or (b) IgA, IgM, IgD, or IgE MM: serum M protein level >=0.5 g/dL or urine M protein level >=200 mg/24 hours; or (c) Light chain MM without measurable disease in serum or urine: serum Ig free light chain (FLC) >=10 mg/dL and abnormal serum Ig kappa lambda FLC ratio
* Participants newly diagnosed and not considered a candidate for high-dose chemotherapy with autologous stem cell transplantation (ASCT) due to being >=65 years old, or in subjects less than (<) 65 years old presence of important comorbid condition(s) likely to have a negative effect on the tolerability of high-dose chemotherapy with ASCT
* Pretreatment clinical laboratory values meeting the following criteria during the Screening Phase
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 4 weeks prior to dosing and the second within 3 days prior to dosing

Exclusion Criteria:

* Participants with diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering MM
* Participant with plasma cell leukemia or other conditions in which Ig (immunoglobulin) M protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Participants who have prior or current systemic therapy or ASCT for MM, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment
* Participants with history of malignancy (other than MM) within 5 years before the date of the first daratumumab administration
* Participants who have radiation therapy within 14 days of the first dose

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) to analyze the safety of daratumumab when combined with lenalidomide and dexamethasone | Cycle 1, Day 1 to Day 28
  Number of Participants With Dose Limiting Toxicity During Cycle 1.

SECONDARY OUTCOMES:
Rate of Complete Response (CR) or Better | Approximately 3.7 years
  CR is Defined as the proportion of Participants achieving CR (including stringent complete response [sCR]) according to the International Myeloma Working Group (IMWG) criteria.
Overall Response Rate (ORR) | Approximately 3.7 years
  ORR is defined as the percentage of participants who achieve CR, Partial Response (PR), VGPR, and sCR according to the IMWG criteria, during or after study treatment.
Very good partial response (VGPR) or better (VGPR, CR, or sCR) | Approximately 3.7 years
  VGPR is serum and urine M-protein detectable by immunofixation but not on electrophoresis or greater than or equal to (>=) 90 pecent (%) reduction in serum M-protein plus urine M-protein level less than (<) 100 milligram(mg)/24 hour (h).
Minimum Observed Serum Concentration (Cmin) | Cycle 1, Cycle 3, Cycle 6, Cycle 12 (each cycle of 28 days), End of Treatment (within 30 days of the last dose), and Follow-Up (8 weeks after the last dose)
  The Cmin is the minimum observed analyte concentration.
Maximum Observed Concentration (Cmax) | Cycle 1, Cycle 3, Cycle 6, Cycle 12 (each cycle of 28 days), End of Treatment (within 30 days of the last dose), and Follow-Up (8 weeks after the last dose)
  The Cmax is the maximum observed analyte concentration.
Immunogenicity of daratumumab | Cycle 1, Cycle 3, Cycle 12 (each cycle of 28 days), End of Treatment (within 30 days of the last dose), and Follow-Up (8 weeks after the last dose)
  Anti-daratumumab antibodies will be evaluated in serum samples collected for all the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (5):
- Japan (5):
  - Hiroshima
  - Kanazawa
  - Nagoya
  - Osaka
  - Shibuya City

REFERENCES:
- [Derived] Takamatsu H, Iida S, Shibayama H, Shibayama K, Yamazaki H, Suzuki K. Daratumumab, lenalidomide, and dexamethasone in Japanese patients with transplant-ineligible newly diagnosed multiple myeloma: a phase 1b study. Int J Hematol. 2020 May;111(5):692-701. doi: 10.1007/s12185-020-02825-w. Epub 2020 Jan 30. PMID 32002821